CLINICAL TRIAL: NCT06558110
Title: Examining the Effect of Internet Use on Exercise Attitudes and Sleep Quality of Students at the Faculty of Health Sciences
Brief Title: Examining the Effect of Internet Use on Exercise Attitudes and Sleep Quality of University Students
Status: Completed | Type: Observational
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Furkan Çakır, Principal Investigator, Istanbul Bilgi University
Other Study IDs: IstanbulBUFC7
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Internet Addiction
Keywords: university students; sleep quality; physical activity
MeSH Terms: conditions — Internet Addiction Disorder; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students: Students of the Faculty of Health Sciences in Istanbul

SUMMARY:
The internet is one of the most critical elements of our age that is rapidly developing and changing. Situations such as the increase in the use of developing and widespread technological products and the addiction of social media application algorithms can negatively affect the health and success of students. Internet addiction among university students can have negative effects on general health parameters and academic success of students. This study will be conducted to determine the effect of internet use on exercise attitudes and sleep quality of foundation university health sciences faculty students. The study is planned to be conducted in the 2024-2025 fall semester and to include at least 1000 students.

DETAILED DESCRIPTION:
The convenience and quick access provided by the internet have made it indispensable for many people. However, the excessive amount of time spent on the internet has led to the phenomenon known as "Internet Addiction." Internet addiction is characterized by an inability to distance oneself from internet use even if desired, spending more time online than initially planned, lying to spend more time on the internet, neglecting responsibilities due to internet use, and experiencing social isolation.

Internet addiction among health sciences students is a significant concern due to its potential impact on general health and academic performance. As the level of internet addiction increases among students, sleep quality and exercise behaviors, which are crucial for health, may be adversely affected. Insufficient, irregular, and poor-quality sleep can lead to sleep disorders, which in turn are significant public health concerns due to their association with incidents like traffic and work accidents. Furthermore, sleep disorders can negatively affect academic success.

Understanding the factors influencing internet addiction behaviors among health sciences students is essential for developing targeted interventions and educational programs to address these issues effectively. Engaging in regular sports and exercise from childhood to adolescence and into old age is crucial for maintaining physical health. It is well known that regular and consistent exercise helps protect against diseases and maintains body weight. Research indicates that regular physical activity can control blood pressure and blood sugar, reduce the risk of colon cancer and coronary heart disease, and prevent musculoskeletal disorders. Regular physical activity has numerous physiological benefits and also positively impacts mental and emotional health.

University students, who are transitioning into adulthood, may experience significant physical, emotional, and cognitive changes. During this period, various factors may cause issues such as poor sleep quality among university students. Sleep quality is defined as feeling refreshed, fit, and ready for a new day upon waking.

Therefore, it is essential to determine the levels of internet addiction and sleep problems among university students, assess their perceptions and attitudes towards physical activity and exercise as part of a healthy lifestyle, and provide proper guidance and encouragement.

This planned study aims to determine the profiles of internet use, exercise attitudes, physical activity status, and sleep quality among health sciences faculty students.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30
* Being willing to participate in the study.
* Being a student at the Faculty of Health Sciences

Exclusion Criteria:

* Being a student other than the Faculty of Health Sciences or at a college
* Refusing to participate in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the research consists of Health Science Faculty students of foundation universities in Istanbul.
Sampling Method: Non-Probability Sample
Enrollment: 1024 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Internet Addiction Scale | Baseline
  The Internet Addiction Scale, which has been adapted to Turkish, will be used. The Internet addiction scale is a 5-point Likert-type scale consisting of 19 items (1= Not Appropriate at All, 2= Somewhat Appropriate, 3= Appropriate, 4= Quite Appropriate, 5= Completely Appropriate). The ceiling score that can be obtained from this scale is 95, and the base score is 19. High scores obtained from the scale indicate that individuals have high levels of internet addiction. According to the reliability analyses of the scale, the internal consistency coefficients of the factors were 0.90 for loss of control, 0.88 for excessive desire to stay online, and 0.92 for negativity in social relationships, and the internal consistency coefficient for the overall scale was determined as 0.85.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline
  The Pittsburgh Sleep Quality Index (PSQI) used to evaluate students' sleep quality is a self-report scale that evaluates sleep quality and sleep disturbance in the last month. It has been shown to have sufficient internal consistency, test-retest reliability and validity. The validity and reliability of the index has been conducted in Turkey and it has been determined that it is suitable for the Turkish society. Cronbach α internal consistency coefficient was determined as 0.80. 18 items are included in the scoring in the evaluation of the PSQI. The PSQI has 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance-conditions affecting sleep, use of sleep-inducing drugs/substances and daytime dysfunction/sleepiness. Total score between 0-4 indicates good sleep quality, and between 5-21 indicates poor sleep quality.
International Physical Activity Questionnaire-Short Form | Baseline
  The International Physical Activity Questionnaire-Short Form was developed to determine the physical activity levels of participants between the ages of 15-65. Validity and reliability studies were conducted in Turkey and test-retest reliability was reported as 0.69. In the evaluation of all activities, the criterion is that each activity is performed for at least 10 minutes at a time. Scoring is done based on the Metabolic Equivalent of Task (MET) value. A score is obtained as "METminutes/week" by multiplying minutes, days and MET values. The physical activity levels of the participants will be classified as physically inactive (<600 MET-min/week), low physical activity level (600-3000 METmin/week) and sufficient physical activity level (beneficial for health) (>3000 METmin/week).
Exercise Benefits/Barriers Scale | Baseline
  The Exercise Benefits/Barriers Scale, is designed to determine people's perceptions of benefits and barriers of exercise. The higher the total score on the scale, the more they perceive the benefits of exercise. The validity and reliability of the scale in Turkey was conducted and the Cronbach alpha coefficient was determined as 0.95. The scale is in Likert format (1: strongly disagree, 2: disagree, 3: agree, 4: strongly agree) and consists of 43 questions in total.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Yorulmaz, Prof., Study Director — Halic University
Locations (1):
- Istanbul Bilgi University, Istanbul, Beyoglu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided